CLINICAL TRIAL: NCT04025034
Title: Deep Lateral Wall Partial Rim-Sparing Orbital Decompression With Ultrasonic Bone Removal for Treatment of Thyroid-Related Orbitopathy
Brief Title: Deep Lateral Wall Partial Rim-Sparing Orbital Decompression for Treatment of Thyroid-Related Orbitopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Hospital del Rio Hortega (Other); The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Enrique Mencia-Gutierrez, M.D., Hospital Universitario 12 de Octubre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLWP-R2019
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Exophthalmos; Orbitopathy, Graves; Surgery
Keywords: Decompression; Thyroid-related; Orbitopathy
MeSH Terms: conditions — Exophthalmos; Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Retrsopective, non-comparative case series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Use of SONOPET(R) to orbital surgery.
  Interventions: Procedure: Orbital decompression with ultrasonic bone removal

INTERVENTIONS:
Procedure: Orbital decompression with ultrasonic bone removal — Deep lateral wall partial rim-sparing decompression for thyroid-related orbitopathy using SONOPET® appears to be safe and effective, reducing the complications associated and damage to neurovascular structures.

SUMMARY:
The described technique of DLW-PRS decompression for TRO using SONOPET(R) appears to be safe and effective, reducing the complications associated with decompressing the orbital floor and medial wall. The mechanical characteristics of this surgical too provide protection to adjacent dura mater and neurovascular structures when working in narrow spaces.

DETAILED DESCRIPTION:
We included in this review patients who had exophthalmos at presentation (using Hertel's exophthalmometer), underwent surgery for rehabilitation of disfiguring exophthalmos and had controlled thyroid function. All patients had a minimum follow up of 6 months. Procedures that potentially might have altered the amount of retroplacement achieved by lateral wall removal, such as fat excision, rim advancement, or decompression into the paranasal sinuses, were not performed. Patients with any history of previous procedures that potentially might have altered exophthalmos measurements were also excluded for the purposes of this study.

SONOPET® Ultrasonic Aspirator. The SONOPET® ultrasonic aspirator, consists of an ultrasonic handpiece that is connected to a base control module. The unit is foot-pedal controlled. The base module houses the controls to regulate the irrigation rate (between 3 and 40 mL/min), aspiration and ultrasound power parameters of the machine. The power setting is expressed as a percentage of that maximum. Aspiration reaches 500 mmHg and the aspiration setting on the machine is also expressed as a percentage of that maximum. The irrigation rate is expressed in milliliters per minute.18 Aspiration occurs through an opening at the distal aspect of the handpiece tip and the irrigation fluid (normal saline at 20°C) flows through a white irrigation sleeve surrounding the handpiece tip. The handpiece oscillates in a nonrotational fashion up to 25,000 times per second with a 0.36 mm width variation. The SONOPET®'s primary mechanism of action is torsional oscillation of a metal bone rasp at 25 kHz. This frequency is ideal for bone removal,22 as the microenvironment created only cuts mineralized tissue, while soft tissues are best cut at frequencies ≥34 kHz.23 The universal handpiece fits multiple interchangeable tips that have varying lengths, sizes, and shapes designed for specific soft tissue or bone removal purposes.22 Different sizes and angles for the cutting surface are also available.

The tip used in this series is a serrated aggressive knife and the superlong payner 360°shape designed for bone fragmentation and removal24 (Figures 1 D, 2 A).

Surgical technique. The procedure was performed with the patient in a supine position under general anesthesia. A single dose of IV dexamethasone (8 mg) and a 1 gr IV cefazoline were given during surgery. After corneal lubrication, the patient was prepped and draped in sterile fashion.

The marked triangle incision was incised (Figure 1, A) and an initial lateral canthotomy was made in a "crow's foot" using a no. 15 Bard-Parker® surgical blade (Becton Dickinson, Hancock, NY, USA) . Dissection was performed in the preseptal plane to provide wide exposure of the rim of the lateral orbital wall(Figure 1, B). The periosteum was incised using a needle-tip monopolar electrocautery and the lateral wall was completely exposed by cutting cautery and periosteal elevators (Figure 1, C). The posterior leaf of the periosteum was mobilized and reflected, along with the temporalis muscle; this minimizes damage to the temporalis muscle during surgery and reduces future temporal hollowing.

ELIGIBILITY:
Inclusion Criteria: Exopthalmos -

Exclusion Criteria: Previous procedures

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Orbital decompression in exophthalmos in treatment of thyroid-related orbitopahty | 33 months
  Decompression with a bone-cutting ultrasonic aspirator that can be customized for variable decompression of the orbit by tailoring the amount of bone removed from each wall.
Change in proptosis | 33 months
  Measured by the difference in Hertel exophthalmometry

SECONDARY OUTCOMES:
Visual acuity | 33 months
  Using Snellen scale, decimal fraction
Lagophthalmos | 33 months
  Presence of lagophthalmos
Eyelid retraction | 33 months
  Measured by upper eyelid margin distance to the corneal reflex and lower eyelid margin distance to the corneal reflex
Keratopathy | 33 months
  Presence of exposure keratopathy

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ugalde-Diez, M.D., Ph.D., Study Director — 12 de Octubre Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Yes
To describe the results of thyroid-related orbitopathy (TRO) treated by ultrasound lateral deep lateral wall bony decompression with partial rim sparing (DLW-PRS)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: A review was carried out, from January 2015 to September 2017, of all patients treated with ultrasound DLW-PRS decompression using a SONOPET® (Striker, Kalamazoo, MI, USA)
Access Criteria: The primary outcome was the change in proptosis (measured by the difference in Hertel exophthalmometry measurements). Other secondary outcomes were changes in visual acuity (VA) (using Snellen scale, decimal fraction), presence of lagophthalmos, eyelid retraction (measured by superior eyelid margin distance to the corneal reflex (MRD1) and inferior eyelid margin distance to the corneal reflex (MRD2)), and presence of exposure-related symptoms and exposure keratopathy.

REFERENCES:
- [Result] Baldeschi L, MacAndie K, Hintschich C, Wakelkamp IM, Prummel MF, Wiersinga WM. The removal of the deep lateral wall in orbital decompression: its contribution to exophthalmos reduction and influence on consecutive diplopia. Am J Ophthalmol. 2005 Oct;140(4):642-7. doi: 10.1016/j.ajo.2005.04.023. Epub 2005 Sep 2. PMID 16140250
- [Result] Paridaens DA, Verhoeff K, Bouwens D, van Den Bosch WA. Transconjunctival orbital decompression in Graves' ophthalmopathy: lateral wall approach ab interno. Br J Ophthalmol. 2000 Jul;84(7):775-81. doi: 10.1136/bjo.84.7.775. PMID 10873993
- [Result] Sivak-Callcott JA, Linberg JV, Patel S. Ultrasonic bone removal with the Sonopet Omni: a new instrument for orbital and lacrimal surgery. Arch Ophthalmol. 2005 Nov;123(11):1595-7. doi: 10.1001/archopht.123.11.1595. PMID 16286624
- [Result] Cho RI, Choe CH, Elner VM. Ultrasonic bone removal versus high-speed burring for lateral orbital decompression: comparison of surgical outcomes for the treatment of thyroid eye disease. Ophthalmic Plast Reconstr Surg. 2010 Mar-Apr;26(2):83-7. doi: 10.1097/IOP.0b013e3181b8e614. PMID 20305505
- [Derived] Bengoa-Gonzalez A, Galindo-Ferreiro A, Mencia-Gutierrez E, Sanchez-Tocino H, Martin-Clavijo A, Lago-Llinas MD. Deep Lateral Wall Partial Rim-Sparing Orbital Decompression with Ultrasonic Bone Removal for Treatment of Thyroid-Related Orbitopathy. J Ophthalmol. 2019 Dec 2;2019:9478512. doi: 10.1155/2019/9478512. eCollection 2019. PMID 31885895
- See also: Navigator — http://microsoftwindows.com
- Available data/document: Informed Consent Form — http://microsoftwindows.com — Navigator